CLINICAL TRIAL: NCT02778516
Title: Sodium-restricted Diets and Symptoms in End Stage Renal Disease: An RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Maya N. Clark-Cutaia, Adjunct Faculty, Lecturer N, University of Pennsylvania
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 819779
Record Dates: First submitted 2015-06-08; First posted 2016-05-20 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: ESRD
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sodium Restriction 1500mg Group (Active Comparator): During the intervention phase of the study, participants will consume iso-caloric diets provided by the CTRC Nutrition Services Metabolic Kitchen at the UPHS. Diets will differ only in sodium content. To ensure accurate calculation of calorie and dietary sodium content for each individual, sodium content from all uneaten foods will be deducted from total daily dietary sodium intake. Total sodium intake will be calculated by CTRC Nutrition Staff and recorded on the data collection sheet after each meal and used in final analyses.
  Interventions: Dietary Supplement: Sodium Restriction
- Sodium Restriction 2400mg Group (Active Comparator): During the intervention phase of the study, participants will consume iso-caloric diets provided by the CTRC Nutrition Services Metabolic Kitchen at the UPHS. Diets will differ only in sodium content. To ensure accurate calculation of calorie and dietary sodium content for each individual, sodium content from all uneaten foods will be deducted from total daily dietary sodium intake. Total sodium intake will be calculated by CTRC Nutrition Staff and recorded on the data collection sheet after each meal and used in final analyses.
  Interventions: Dietary Supplement: Sodium Restriction
- Control Group (No Intervention): During the intervention phase of the study, participants will consume iso-caloric diets provided by the CTRC Nutrition Services Metabolic Kitchen at the UPHS. Diets will differ only in sodium content. To ensure accurate calculation of calorie and dietary sodium content for each individual, sodium content from all uneaten foods will be deducted from total daily dietary sodium intake. Total sodium intake will be calculated by CTRC Nutrition Staff and recorded on the data collection sheet after each meal and used in final analyses.

INTERVENTIONS:
Dietary Supplement: Sodium Restriction
  Arms: Sodium Restriction 1500mg Group; Sodium Restriction 2400mg Group

SUMMARY:
Dietary sodium intake independently increases the risk of mortality in end stage renal disease (ESRD). It plays a significant role in hypertension, hypervolemia, and left ventricular hypertrophy (LVH), and blunts the effectiveness of hypertensive agents. In addition, the hypervolemia associated with excessive dietary sodium intake results in the need for more intense fluid removal during dialysis (ultrafiltration), resulting in symptoms such as pain, cramps, hypotension, nausea, and vomiting during hemodialysis (HD) treatment sessions. Although sodium restriction is a universal recommendation for ESRD management, the National Kidney Foundation (NKF) recommendation of 2400 mg/day is consensus-based per the Dietary Approaches to Stop Hypertension (DASH) studies, not an evidence-based recommendation from data derived from a dialysis population. In addition, The Dietary Guidelines for Americans 2010, recommend further restriction of dietary sodium intake to 1500 mg per day for persons with hypertension and/or kidney disease, middle-aged and older adults, and African Americans, though there is also little empiric evidence to support this recommendation in the general population and none in the dialysis population. Therefore, it remains to be demonstrated that a diet with such sodium restrictions is attainable, sustainable, safe or beneficial. The investigators propose a double blind randomized controlled design investigation to examine the feasibility of assessing the effects of three levels of sodium intake (ambient, 2400 mg/d, 1500 mg/d) on the hemodialysis (HD) participant symptom profile, and to compare the effect of hemodialysis-specific variables on participant symptom profile during dialysis as well as to explore the role of body fluid composition using bioimpedance (BIA) measurements among the three sodium-restricted groups as a marker of sodium restriction efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. persons ≥ 21 years of age
2. who have the ability to read and write,
3. who are undergoing maintenance HD
4. who are on therapy for at least 3 months.

Exclusion Criteria:

1. unable to read or write
2. non-English speaking
3. intend to move out of the area or change HD centers within 6 months
4. have terminal illness or life expectancy of less than 12 months,
5. plan to receive a living donor transplant in the study period, have cognitive impairment
6. are unable to provide informed consent
7. have heart Failure Class III or IV
8. have an internal defibrillator or pacemaker, and/or are pregnant.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Interdialytic Weight Gain | 5 days
  IDWG is defined as the difference in weight in kilograms between measurement at time 1 (immediately following HD) and time 2 (immediately prior to the next HD session).4 Weights will be obtained in the aforementioned fashion in the CTRC, and calculated by the CTRC nursing core staff. The PI will train CTRC personnel on IDWG calculations.
Palliative Care Outcomes Scale-Renal | 3-5 days
  The POS is a survey used to measure health related QOL in the short term.68, 69 It reviews the symptoms listed in the KDQOL-36, however, the respondent refers to these symptoms in the short-term, the last three days
Body Composition | 5 days
  Body composition will be measured with bioimpedance spectroscopy (BIS; ImpediMed® Imp_ SFB7, ImpediMed Limited, Queensland, Australia). Measurements include TBW, ECF, and ICF (in liters). We will take three consecutive measurements on the external surface of the skin by placing electrodes on the right hand and right foot. BIS has been shown good correlation with biochemical markers, such as the gold standard tracers methods (R2=0.93) when measuring ECF62, 63, but may have better clinical application due to its ease of use, reproducibility, and the fact that biochemical markers are costly and require vast amounts of training to perform, limiting the availability of analysis centers.

SECONDARY OUTCOMES:
Blood Pressure. | 5 days
  An oscillometric device, fitted with an appropriate cuff, will be used to measure mean systolic and mean diastolic pressure in the CTRC in accordance with World Health Organization guidelines.61 These same guidelines will be used by DaVita Dialysis center staff during blood pressure measurements. DaVita nursing will be trained by the PI to ensure adherence to blood pressure measurement protocols

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania School of Nursing, Philadelphia, Pennsylvania, United States